CLINICAL TRIAL: NCT07190456
Title: Kinesiophophia or Task-specific Fear of Movement? What Are we Talking About in Patients Post Anterior Cruciate Ligament Reconstruction?
Brief Title: Kinesiophobia vs. Task-Specific Fear: Defining Movement-Related Fear in ACL Reconstruction Patients
Acronym: Ki-TASK-ACLR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1476
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: ACL Reconstruction
Keywords: Motor behavior; gait complexity; Autonomic Nervous System; Heart Rate Variability; Skin Conductance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neutral images (Sham Comparator): The patient will have to walk on a treadmill at their preferential walking speed for 10 minutes while visualizing neutral images (landscapes, monuments...)
  Interventions: Other: Exposure to neutral images visualization
- Nocive images (Experimental): The patient will have to walk on a treadmill at their preferential walking speed for 10 minutes while visualizing images interpreted as nocive (cutting, jumping, contact...)
  Interventions: Other: Exposure to nocive images visualisation
- Antecipation feared movement (Experimental): Before the start of the experimental condition, the patient will be asked to think about their willingness to perform the first movement visualised in the video, while a researcher places a jumping platform inside the laboratory.
  During the test, the patient will have to walk on a treadmill at their preferred speed for 10 minutes, while watching a video showing a drop jump followed by images interpreted as nocive for the rest of the time.
  Interventions: Other: Exposure to anticipated realisation of a feared movement

INTERVENTIONS:
Other: Exposure to neutral images visualization — The patient will have to walk on a treadmill at their preferential walking speed for 10 minutes while visualizing neutral images (landscapes, monuments...)
  Arms: Neutral images
Other: Exposure to nocive images visualisation — The patient will have to walk on a treadmill at their preferential walking speed for 10 minutes while visualizing images interpreted as nocive (cutting, jumping, contact...)
  Arms: Nocive images
Other: Exposure to anticipated realisation of a feared movement — Before the start of the experimental condition, the patient will be asked to think about their willingness to perform the first movement visualised in the video, while a researcher places a jumping platform inside the laboratory. During the test, the patient will have to walk on a treadmill at their preferred speed for 10 minutes, while watching a video showing a drop jump followed by images interpreted as nocive for the rest of the time.
  Arms: Antecipation feared movement

SUMMARY:
Kinesiophobia, defined as an excessive and irrational fear of physical movement due to perceived vulnerability to injury, has gained significant attention in clinical and scientific communities. This condition can act as a barrier to physical activity, negatively impacting patients' disability, quality of life, and the implementation of rehabilitation programs. It is particularly prevalent after anterior cruciate ligament reconstruction (ACLR), affecting physical function, return to sport rates, and patient performance.

While the Tampa Scale for Kinesiophobia (TSK) is considered a gold standard for assessing kinesiophobia, recent studies have raised concerns about its validity, especially in ACLR patients. The TSK may not adequately capture fear of specific sports activities, which is more common in ACLR patients than a general phobia of movement. Some researchers argue for an assessment approach similar to that used for pain experiences, emphasizing the subjective nature of fear.

Based on the specific phobia model, assessing kinesiophobia in the presence of a trigger, such as visualizing or confronting the movement associated with the injury, may be more relevant. This approach is supported by evidence showing that sports situations evoking the greatest fear after ACLR are cutting, jumping, and contact. Further research is needed to investigate alternative methodologies for assessing fear of movement in ACLR patients, considering the prevalence and repercussions of kinesiophobia in this population.

The objectives of this study are threefold:

* To compare the magnitude of kinesiophobia through the TSK, the subjective feeling of fear when visualising feared movements, and the subjective feeling of fear in anticipation of the feared situation.
* Evaluate the impact of focusing on feared activities on motor behavior and Autonomic Nervous System (ANS) markers.
* To assess the relation between the three methods of assessing fear of movement and indicators of motor behaviour, ANS activity, fear-avoidance beliefs, anxiety, avoidance behaviour, and physical function.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their informed consent and signed the consent form.
* The patient must have enough comprehension of the Portuguese language to complete the written questionnaires.
* The patient must have suffered an ACL injury, with or without a history of concomitant meniscal pathology, while playing or training for sport (recreational or organized).
* The patient must have undergone anterior cruciate ligament reconstruction surgery.
* The patient must be between 18 and 35 years old.
* The patient must still be under medical care/rehabilitation due to the ACL injury.
* The patient must have started jump landing tasks.

Exclusion Criteria:

* The subject has a history of repeated ACLR.
* The subject has not injured the ACL while playing sports.
* The subject presents a concurrent psychiatric disorder
* The subject has a history of heart disease and/or peripheral vascular disease and/or metabolic disease and/or Raynaud´s Syndrome.
* The subject is taking any medications known to affect heart rate or blood pressure
* The subject is currently a smoker.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Fractal scaling exponent (α) | Day 0 (during intervention)
  The fractal scaling exponent quantifies the complexity of a physiological signal and detects the presence of statistical persistence in a given time series. This parameter is calculated using Detrended Fluctuation Analysis (DFA) from each time series (stride time and stride length).
Heart rate variability | Day 0 (during intervention)
  The R-R intervals will be derived from beat-to-beat blood pressure pulse intervals using finger plethysmography (Finapres® Nova, Amsterdam, Netherlands), at rest and during the gait trials. Finger plethysmography-derived peak-to-peak intervals are highly correlated with ECG R-R intervals, with similar variability. The upstroke is determined using the pressure signal with a resolution of 2 ms, and the interval between the two consecutive upstrokes is measured. In the frequency domain, the two primary components are low-frequency (LF; 0.04-0.15 Hz) and high-frequency (HF; 0.15-0.40 Hz) spectra. Heart rate variability measures provide information primarily on vagal modulation with the LF power spectrum reflecting both sympathetic and parasympathetic modulation and HF acting as a surrogate marker of parasympathetic modulation of the R-R intervals. The LF/HF ratio is used to indicate sympathovagal dominance.
Skin conductance | Day 0 (during intervention)
  The skin conductance response (SCR) of the patients will be measured while they are exposed to the stimuli of the three experimental conditions. The SCR is an indicator of physiological arousal and is measured by detecting changes in the electrical conductance of the skin, which varies with the activity of the sweat glands. This assessment aims to understand the response of the patient's autonomic nervous system to the experimental conditions.
Blood pressure variability | Day 0 (during intervention)
  Systolic and diastolic blood pressure values will be derived from beat-to-beat blood pressure recordings using finger plethysmography during all gait trials. Finger plethysmography-derived systolic and diastolic blood pressure signals are recorded with high precision and beat-to-beat variability in blood pressure is calculated with a resolution of 2 ms.
  The variability is assessed by measuring the intervals between consecutive systolic upstrokes in the blood pressure waveform. BPV is analyzed by decomposing the signal into two primary components: low-frequency (LF; 0.04-0.15 Hz) and high-frequency (HF; 0.15-0.40 Hz) spectra. Blood pressure variability in the LF range reflects sympathetic modulation of vascular tone and arterial baroreflex sensitivity, while HF variability is often associated with respiratory influences and parasympathetic activity. The LF/HF ratio is used as an indicator of the balance between sympathetic and parasympathetic contributions to blood pressure regulation.

SECONDARY OUTCOMES:
Physical Function in Sports and Leisure Activities subscale of the Knee Injury and Osteoarthritis Outcome Score (KOOS-Sport/Rec) | Day 0 (Before experiment)
  The KOOS is a self-reported measure that allows assessing a broad spectrum of subjects with knee injuries and OA, concerning pain and other symptoms, daily life function, sport and recreation, and knee-related quality of life. It consists of five sub-scales which are scored separately: pain (nine items); symptoms (seven items); function in ADL (17 items); Function in Sport and Recreation (five items); and Quality of Life (four items). The items are scored on a 5-point Likert scale ranging from 0 (no problems) to 4 (extreme problems). We will use the "Function in Sport and Leisure" subscale of the Portuguese version of the KOOS, for which total scores can range between 0 and 25 points, where zero represents extreme knee problems and 25 represents absence of knee problems.
Physical Activity subscale of the Fear-Avoidance Beliefs Questionnaire (FABQ-PA) | Day 0 (Before experiment)
  Fear-avoidance beliefs will be assessed using the Portuguese version of the FABQ. The original questionnaire was developed for subjects with chronic low back pain and consists of 16 items divided into two subscales, the FABQ-Physical Activity (FABQ-PA) and the FABQ-Work. The Portuguese version consists of 15 items, as item 8 ("I made a request for work compensation because of my pain") of the original scale was removed for being problematic. The subscale FABQ-PA of the Portuguese version consists of 5 items and the FABQ-work subscale consists of 10 items. In this study, we will use the FABQ-PA subscale specific to the knee, in which "back" will be replaced by "knee" as previously proposed in the literature. The 5 items of the FABQ-PA are scored on a 6-point Likert scale, except item 1 which is not quoted. The total score for the sub-scale can therefore range between 0 and 24 points. Higher scores on the FABQ indicate higher levels of fear-avoidance beliefs.
Tampa Scale for Kinesiophobia 13 items version (TSK-13) | Day 0 (Before experiment)
  To assess kinesiophobia, the Portuguese version of the Tampa Scale for Kinesiophobia (TSK-PT), consisting of 13 items, will be used. The individual items are scored on a 4-point Likert scale (1 to 4), where 1 corresponds to "totally disagree" and 4 corresponds to "totally agree". The total score on the scale ranges between 13 and 52, with higher scores indicating higher levels of kinesiophobia.
Hospital Anxiety and Depression Scale (HADS) | Day 0 (Before experiment)
  HADS is a screening instrument for anxiety and depression that helps to recognize the emotional components of physical illness. Structurally, it consists of two subscales, one assessing anxiety (HADS-A) and the other assessing depression (HADS-D). Each subscale contains 7 items, which are scored from 0 to 3 on a Likert scale. The total scores for each subscale range between 0 and 24 points.
  We will use the HADS-A of the Portuguese version of the scale. The HADS-A contains items 1,3,5,7,9,11 and 13 of the scale, all of which score inversely except for items 7 and 9. According to the HADS manual a score between 0 and 7 is considered "normal", between 8 and 10 indicates "mild" anxiety, between 11 and 14 "moderate" and between 15 and 21 "severe" anxiety. Other authors propose a cut-off value of 8/9 points.
Subjective feeling of fear (SFoM) | Day 0 : After walking with visualization of neutral images; after walking with visualization of feared movements; after walking with visualization of feared movement and in the anticipation of realizing a feared movement.
  Numerical Rating Scale [0;100]
Avoidance behaviour related to specific feared activities | Day 0: after walking with visualization of feared movement and in anticipation of realizing a feared movement.
  Participants will be asked to rate their agreement on a 0 to 100 numerical rating scale, with zero representing "totally disagree" and 100 representing "totally agree", with the following statement: "Because I am afraid of pain and/or re-injury I prefer to avoid jumping"
Coefficient of Variation (CV) | Day 0 (during intervention)
  CV is a common linear measure that translates the amount of variability within the signal and is calculated through the standard deviation normalised to the mean from each time series (stride time and stride length).

OTHER OUTCOMES:
Subjective level of immersion | Day 0: At the end of the experimental conditions
  Participants will be invited to rate their agreement with the statement "Somehow I felt that the visual aspects involved me". The statement was adapted from item 9 of the Portuguese version of the Presence Questionnaire. This questionnaire is normally used in virtual reality studies to characterize the magnitude of the sensation of presence. The answer is scored on a 5-ponint Likert scale ranging from 0 (totally disagree) to 5 (completely agree).

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Clínica de Fisioterapia Egas Moniz, Caparica, Almada
  - Egas Moniz School of Health & Science, Almada, Monte Da Caparica

IPD SHARING:
Plan to Share IPD: No